CLINICAL TRIAL: NCT05994885
Title: Prognostic Potentials of E-cadherin and Total Antioxidant Capacity in Gingival Crevicular Fluid of Moderately Deep Periodontal Pockets Treated With Nonsurgical Periodontal Therapy
Brief Title: Evaluation of Prognostic Potentials of Gingival Crevicular Fluid E-cadherin and Total Antioxidant Capacity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ali A Abdulkareem (Other)
Responsible Party: Sponsor-Investigator, Ali A Abdulkareem, Assistant Professor, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 747622
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients with periodontitis, of any stage, having periodontal pockets of a moderate depth (4 to 6 mm) treated with nonsurgical periodontal therapy.
Masking Description: The care provider is not aware about clinical parameters and biochemical analysis of GCF (E-cadherin and total antioxidant capacity).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Root surface debridement (Other): Periodontal pockets with PPD of 4 to 6mm are treated with root surface debridement only and assessed after 3 months for success/failure of treatment.
  Interventions: Procedure: Root surface debridement

INTERVENTIONS:
Procedure: Root surface debridement — the included patients will undergo full-mouth supra- and subgingival debridement by using ultrasonic device and manual instrumentation at baseline. This is followed, after 1 week, by performing root surface debridement for all pockets with PPD = 4-6 mm for each patient. All patients will be instructed to brush their teeth twice daily and will be supplied with the same type of tooth paste and toothbrush, with suitable interdental aids.

SUMMARY:
Ability to anticipate the outcomes of periodontal therapy at baseline visit is crucial to outline and customize a treatment plan with predictable outcomes and cost-effectiveness. Presence of diverse range of health/disease-associated molecules in oral environment that reflect health and disease, together with clinical parameters, is an appealing approach to use them as biomarkers to diagnose, predict, and monitor periodontal disease. Among these proteins are E-cad and TAC which available evidence indicate that their concentrations in oral biofluids increase remarkably during periodontitis as compared to healthy periodontium.

DETAILED DESCRIPTION:
Loss of attachment and formation of periodontal pockets are hallmarks of periodontitis. The treatment approach is either by nonsurgical or surgical periodontal therapy or a combination of both depending on the severity of the case. In general, sites with moderately deep pockets (4 to 6 mm) are responding favorably to nonsurgical periodontal therapy (NSPT). Nevertheless, some sites exhibit persistent pockets even with multiple treatment sessions which could be attributed to the presence of tissue invaders or aberrant immune response that impede healing process.

Prediction of treatment outcomes based on clinical data is limited and sometimes lacking accuracy. Use of biomarkers that can be non-invasively collected from oral fluids e.g., gingival crevicular fluid (GCF) as diagnostic/predictive tools has gained attention in the last decade. For instance, E-Cadherin (E-cad) and total antioxidant capacity (TAC) are associated with periodontitis. E-cad is a transmembrane glycoprotein that is a key mediator of stable cell-cell adhesion of epithelial cells. E-cadherin-based adherens junctions specialized cell structures that mediate cell-cell adhesion and regulate cytoskeleton reorganization forming a continuous, linear circumferential belt (zonula adherens) around the apical part of the cell. While TAC, defined as the moles of oxidants neutralized by one liter of solution, is a biomarker measuring the antioxidant potential of body fluids.

Available evidence indicates that the concentration of both molecules are substantially increased with increasing severity of periodontitis and vice versa in periodontal health. This suggests the potential of GCF-E-cad and TAC to predict the prognosis following NSPT.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy adult patients (> 18 years).
* Periodontitis (interdental clinical attachment loss (CAL) detectable at ≥2 non-adjacent teeth, or buccal/oral CAL of ≥3mm with pocketing of >3mm is detectable at ≥2 teeth). All patients should exhibit generalized periodontitis with pockets of PPD = 4 to 6 mm of any stage, unstable, and grade A to C. Only maxillary teeth with single root will be included.

Exclusion Criteria:

* Consumption of antibiotics or periodontal treatment 3-months prior to the study.
* Pregnancy and lactation.
* Smoker.
* History of systemic disease e.g., diabetes mellitus.
* Patients currently recruited in other trials.
* Patients not willing to consent.
* Periodontal pockets ≥ 7mm, active caries, endodontic problem.
* Multi-rooted teeth will be also considered as exclusion reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth | Baseline, 1 week, then 1 month and 3 months after treatment
  Linear distance, in mm, measured from the gingival margin to the base of periodontal pocket or sulcus.

SECONDARY OUTCOMES:
Clinical attachment loss | Baseline, 1 week, then 1 month and 3 months after treatment
  Linear distance, in mm, measured from the cementoenamel junction to the base of periodontal pocket or sulcus.
Bleeding on probing | Baseline, 1 week, then 1 month and 3 months after treatment
  Presence or absence of bleeding is detected after 30 seconds of inserting periodontal probe to the depth of periodontal pocket/sulcus
Gingival crevicular fluid E-cadherin | Baseline, 1 month and 3 months after treatment
  Level of E-cadherin in GCF collected from periodontal pockets is determined by biochemical analysis
Total antioxidant capacity | Baseline, 1 month and 3 months after treatment
  Level of TAC in GCF collected from periodontal pockets is determined by biochemical analysis

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry/ University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No